CLINICAL TRIAL: NCT06200766
Title: A Multicenter, Randomized, Double-blind, Three-arm, Parallel Clinical Endpoint Bioequivalence Study of Monometasone Furoate Nasal Spray in Patients With Seasonal Allergic Rhinitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zheng Liu ENT (Other)
Collaborators: Zhejiang Xianju Pharma Tech. Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Zheng Liu ENT, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJYY-02
Record Dates: First submitted 2023-09-04; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Momethasone furoate nasal spray (trade name: Yiqing®/ Yiqing®) (Experimental): Dosage form: nasal spray Specification: 60 press per bottle, 50 µ g of mometasone furoate, drug concentration: 0.05% (g / g) Route of administration: nasal injection Storage: 2℃ ~25℃ storage Manufacturer: Zhejiang Xianju Pharmaceutical Co., Ltd Specific administration method: 2 snap (50 µ g per snap), total 4 snap (total 200 µ g), 1 time / day.
  Interventions: Drug: Mometasone furoate as a nasal spray
- Momethasone furoate nasal spray (trade name: Nasonex ®/ Nasonex ®) (Active Comparator): Dosage form: nasal spray Specification: 60 press per bottle, 50 µ g of mometasone furoate, drug concentration: 0.05% (g / g) Route of administration: nasal injection Storage: 2℃ ~25℃ storage Holder manufacturer: MSD Belgium BVBA / SPRL Specific administration method: 2 presses (50 per side nostril µ g per snap), total 4 presses (total 200 µ g), One time / day
  Interventions: Drug: Mometasone furoate as a nasal spray
- placebo (Placebo Comparator): Dosage form: nasal spray Specification: 60 press per bottle Route of administration: nasal injection Storage: 2℃ ~25℃ storage Manufacturer: Zhejiang Xianju Pharmaceutical Co., Ltd Specific administration method: 2 presses (50 per side nostril µ g per snap), total 4 presses (total 200 µ g), One time / day
  Interventions: Drug: Mometasone furoate as a nasal spray

INTERVENTIONS:
Drug: Mometasone furoate as a nasal spray — Subjects received 2 presses in each side nostrils at the same time point (± 1h).

SUMMARY:
Taking the mamsonic acid nasal spray held by Zhejiang Xianxian Pharmaceutical Technology Co., Ltd. as the test agent,Bannicate nose spray (product name: inside: insideSchuro®) is a reference preparation. Among the seasonal allergic rhinitis patients, through comparative clinical end, evaluation.The biological equivalent of the two types of branic acid Miimone pine nose spray agent. Observe the test agent and reference preparation in the season.Safety in patients with sexual allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged from 18 to 65 (including boundary value) or non-pregnant or nonlactating women shall agree.

   Appropriate contraceptive measures during the trial (see Appendix 1 for specific measures);
2. Moderate to severe seasonal allergic rhinitis patients, 1 year past history (including the main complaint), diagnosis based on reference to the diagnosis and treatment guidelines of allergic rhinitis (2022, revised), random there are one or more allergens tested positive, approved skin prick test (SPT), serum specific IgE in any allergen test results. If the allergen test report can be provided within 12 months, there is no need to repeat the item;
3. The 12-h total reactive nasal symptom score (rTNSS) assessed during the screening period (Visit 1) was 6 (out of 12), and the nasal congestion score was 2;
4. Prior to the start of the trial, the subjects voluntarily signed the informed consent form approved by the ethics committee;
5. At screening (Visit 1), the subjects could master the correct nasal spray administration method and score the nasal symptoms as required by the protocol.

Exclusion Criteria:

1. Allergic to ometasone furoate or its excipients, or have been shown to be ineffective against ometasone furroate or other glucocorticoids; 2. Having any clinically significant serious medical history or illness that the investigator considers affects subject safety or the conduct of the trial; 3. Severe liver and renal diseases, or abnormal liver and renal function tests with clinical significance (ALT, AST> 1.5 times of normal, times, or TBIL> 1.5 times the upper limit of normal value with any AST, or Cre> 1.2 times the upper limit of normal); 4. Screening of alcohol addicts or drug users in the first 2 years (Visit 1); 5. Select (Visit 1) for nasal trauma who had sinus surgery or incomplete healing within 3 months; 6. Those who have participated in other drug clinical trials and used study drugs within 3 months prior to screening (Visit 1); 7. Those who were vaccinated within 7 days prior to screening (Visit 1) or who are scheduled to be vaccinated during the trial; 8. Presof glaucoma, cataract, ocular herpes simplex, infectious conjunctivitis or other eye infections during screening (Visit 1); 9. Local or systemic fungal, bacterial, viral or parasitic infection with active or inactive pulmonary TB infection at the screening (Visit 1), not cured and still requiring continuous treatment, the subject may be at risk of discomfort or affect the judgment of the test results; 10. Patients with asthma requiring long-term treatment (occasional acute asthma, or mild, exercise-induced asthma, unmedicated or limited to inhaled short-acting β receptor agonists during the trial (patients with a maximum of 8 doses per day can be included)); 11. Screening period or randomized anterior nasal examination results judged by the investigator of nasal diseases or symptoms / signs that may affect the intranasal drug deposition, such as acute or chronic sinusitis, chronic purulent symptoms or signs of the postnasal drip, drug rhinitis, significant nasal polyps, other clinically significant respiratory tract malformations / nasal structure abnormalities, significant nasal trauma (e. g., nasal penetration injury), or significant nasal septum deviation; 12. Patients with any nasal mucosa erosion, septal ulcer or septal perforation during screening or before randomization; 13. The following drugs and / or patients were used during the 7 half-lives before the lead-in period (see Appendix 2): vasoconstrictors (3 days), strong sedative (3 days), antihistamine (3-10 days), decongestants (3 days), leukotriene receptor antagonists (7 days), anticholines (7 days), sweet acids (14 days), systemic antibiotics (14 days), ocular mast cell stabilizers (14 days), monoamine oxidase inhibitors (14 days), tricyclic antidepressants (14 days), potent CYP3A4 Induction / inhibitor (14 days), anti-allergic Chinese herbs (14 days), Corticosteroids (14-30 days), immunotherapy (60-120 days), etc.; 14. planned use of the following drugs or / and treatment during the trial: a. potent CYP3A4 induction / inhibitor; b. Chronic or intermittent use of corticosteroids (except investigational drugs); c. antihistamines (except rescue drugs under protocol); d. leukotriene receptor antagonist; e. mast cell membrane stabilizer; f. [] systemic or intranasal decongestant; g. anticholinic; h. immunosuppresant; i. anti-allergic herbal / Chinese patent / health products; j. anti-IgE antibody (such as Omajumab for injection); k. nasal irrigation agent (including saline); 15. Those who plan to travel for 2 consecutive days or more than 3 days during the trial; 16. Any situation that may affect the subject's informed consent or follow the trial protocol (including compliance with the visit schedule or the diary card or questionnaire, etc.), or that the subject's participation in the trial may affect the trial results or their own safety

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the mean rTNSS versus baseline rTNSS | 4 weeks
  The rTNSS (Reflective Total Nasal Symptom Score) is a scale used to measure nasal symptom severity based on how the patient felt during the previous 12 hours. It is measured on a scale ranging from 0 to 12. Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.

SECONDARY OUTCOMES:
Change in the iTNSS mean from the baseline iTNSS mean during the treatment period. | 4 weeks
  The iTNSS (Instantaneous Total Nasal Symptom Score) is a scale used to measure nasal symptom severity based on how the patient was feeling just before taking each dose of study medication. It is measured on a scale ranging from 0 to 12. Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.

OTHER OUTCOMES:
Number and percentage of patients treated with antihistamine loratadine tablets during the treatment period. | 4 weeks
  The effectiveness of the experimental administration tends to decrease as the frequency of remedial administration increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hosptial affiliated to Tongji Medical college of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No